CLINICAL TRIAL: NCT07249229
Title: Investigating the Effect of Oral L-Carnitine on Inflammatory and Nutritional Factors in Patients With Advanced Kidney Failure Undergoing Chronic Hemodialysis
Brief Title: Oral L-carnitine and Inflammatory and Nutritional Biomarkers in Maintenance Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Darya Chamani (Other)
Responsible Party: Sponsor-Investigator, Darya Chamani, Pharm.D., Principal Investigator, Tehran Islamic Azad University of Medical Sciences
Organization: Tehran Islamic Azad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LC-HD-IAU-2020
Record Dates: First submitted 2025-10-01; First posted 2025-11-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: End-stage Renal Disease (ESRD); Hemodialysis
Keywords: L-carnitine; Hemodialysis; End-stage renal disease; Inflammation; Malnutrition; hs-CRP; Albumin; Ferritin; Lipid profile
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Malnutrition | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-carnitine Group (Experimental): Patients received oral L-carnitine solution (1 g), administered three times per week immediately after each hemodialysis session for 3 months.
  Interventions: Drug: L-carnitine 1000 Mg
- Placebo Group (Placebo Comparator): Patients received placebo solution (distilled water and sodium saccharin), identical in appearance, packaging, and labeling to the active formulation, administered three times per week immediately after each hemodialysis session for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-carnitine 1000 Mg — Participants assigned to the intervention arm received L-carnitine oral solution (1 g) administered three times per week immediately after each hemodialysis session for a total duration of 3 months.
  The oral solution was provided in identical packaging and labeling as placebo to ensure double blinding.
  Arms: L-carnitine Group
Drug: Placebo — Participants assigned to the placebo arm received an oral placebo solution consisting of distilled water and sodium saccharin, three times weekly immediately post-hemodialysis for 3 months, matched to the active formulation in appearance, packaging, and labeling.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to evaluate whether oral L-carnitine supplementation helps reduce inflammation and improve nutritional status in patients with end-stage kidney disease who are undergoing long-term hemodialysis.

A total of 50 participants will be randomly assigned to receive either:

* Oral L-carnitine solution (1 g, three times per week after dialysis), or
* A placebo solution that looks and tastes the same but does not contain L-carnitine.

The study will last for three months. Researchers will assess changes in:

* Inflammatory markers (high-sensitivity C-reactive protein, hs-CRP)
* Nutritional markers (serum albumin, ferritin)
* Blood lipid profile (cholesterol, LDL, HDL, triglycerides)

The findings from this study are expected to provide insights into the potential clinical benefits of oral L-carnitine supplementation in maintenance hemodialysis patients.

DETAILED DESCRIPTION:
This randomized, quadruple-blind, placebo-controlled clinical trial is designed to investigate the effect of oral L-carnitine supplementation on inflammatory and nutritional parameters in patients with end-stage renal disease (ESRD) undergoing chronic hemodialysis (HD).

Study Design and Participants:

The study is conducted at the dialysis departments of Bu Ali Hospital and Partian Clinic in Tehran. Eligible participants are adults (≥18 years) who have been on maintenance HD for at least 6 months, are clinically stable for at least 3 months, and are able to provide informed consent. Patients are excluded if they have a recent infection, malignancy, severe liver disease, uncontrolled comorbidities, or have used anti-inflammatory or lipid-lowering drugs within the previous 3 months.

Randomization and Intervention:

Fifty participants are randomized into two groups. The intervention group receives oral L-carnitine solution (1 g, three times per week after dialysis, produced by Bonyan Salamat Kasra Company). The control group receives a placebo solution (distilled water with sodium saccharin) identical in appearance and packaging. Randomization is computer-generated and allocation is concealed.

Endpoints:

The primary outcome measure is the change in high-sensitivity C-reactive protein (hs-CRP) after three months of intervention. Secondary outcome measures include changes in serum albumin, ferritin, triglycerides, total cholesterol, HDL, and LDL.

This study is intended to help determine whether oral L-carnitine supplementation can improve inflammation, nutritional status, and lipid metabolism in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* On maintenance hemodialysis for at least 6 months
* Clinically stable for ≥ 3 months
* No hospitalization in the preceding 3 months
* Willingness to provide written informed consent and comply with study procedures

Exclusion Criteria:

* Use of statins, erythropoietin, corticosteroids, NSAIDs, or other anti-inflammatory/lipid-lowering agents within the previous 3 months
* Active infection, inflammatory disease, malignancy, or severe hepatic dysfunction
* Pregnancy or breastfeeding
* Participation in another clinical trial within the preceding 3 months
* Uncontrolled comorbidities (e.g., uncontrolled diabetes or hypertension)
* Acute cardiovascular events within the past 6 months
* Planned kidney transplantation during the study period
* Anticipated poor compliance
* Use of medications that could affect inflammatory or lipid parameters
* History of hypersensitivity to L-carnitine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
hs-CRP levels (high sensitivity C-reactive protein) | Baseline and at 3 months after the start of intervention
  Change in serum hs-CRP levels from baseline to 3 months of treatment. hs-CRP will be measured to evaluate systemic inflammation and assess the anti-inflammatory effect of oral L-carnitine supplementation compared with placebo in patients undergoing hemodialysis

SECONDARY OUTCOMES:
Lipid profile (total cholesterol, LDL, HDL, triglycerides) | Baseline and at 3 months after the start of intervention
  Change in lipid profile parameters from baseline to 3 months to assess metabolic impact of L-carnitine
Ferritin levels | Baseline and at 3 months after the start of intervention
  Change in serum ferritin levels from baseline to 3 months as a marker of iron status and inflammation
Serum albumin levels | Baseline and at 3 months after the start of intervention
  Change in serum albumin concentration from baseline to 3 months as an indicator of nutritional status

CONTACTS AND LOCATIONS:
Locations (1):
- Bu Ali Hospital, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient privacy concerns, ethical considerations, and institutional restrictions. Only aggregated results will be published in peer-reviewed journals